CLINICAL TRIAL: NCT04397120
Title: Comprehensive Analysis of Multilevel Factors Affecting Adenoma Detection Rates of Screening Colonoscopy
Brief Title: The Factors Affecting ADR of Screening Colonoscopy
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: CADR-HuY-2005
Record Dates: First submitted 2020-05-16; First posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Adenoma Detection Rate; Colonoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to assess the impact of multilevel factors on the quality of screening colonoscopy, reflected mainly by adenoma detection rate (ADR).

DETAILED DESCRIPTION:
The subjects will include patients who need to screening colonoscopies by 21 endoscopists between January 2019 and December 2019 were retrospectively enrolled in this unit. Multilevel factors, including patient-, proceduralist-, and procedure-level characteristics were analyzed for the relationship with ADR.

ELIGIBILITY:
Inclusion Criteria:

* Patients were retrospectively included in this study if they had undergone a completed colonoscopy.

Exclusion Criteria:

* prior colonoscopy within 3 years;
* medical history of inflammatory bowel disease (IBD), CRC, or abdominal surgery;
* fair or poor quality of bowel preparation (fair quality: some semisolid stool that could be suctioned or washed away but >90% of mucosal surface seen; poor quality: semisolid stool that could not be suctioned or washed away with <90% of mucosal surface seen);
* failure in cecal intubation;
* withdrawal time without removing<6 min.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Endoscopy Department of a university Hospital
Sampling Method: Non-Probability Sample
Enrollment: 13495 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate | After histopathologically examined, reviewed, and confirmed, an average of 7 days.
  the proportion of colonoscopies in which at least one adenoma was detected

CONTACTS AND LOCATIONS:
Overall Officials: Bin Lu, M.D., Principal Investigator — First Affiliated Hospital of Zhejiang Chinese Medical University
Locations (1):
- First Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data sharing will be consider after study